CLINICAL TRIAL: NCT02248116
Title: An Open-label Multicentre, Follow-up Trial to Assess the Long-term Safety and Tolerability of Oral Administration of Talsaclidine 24 mg Tid in Patients With Mild to Moderate Dementia of the Alzheimer Type
Brief Title: Follow-up Trial to Assess the Long-term Safety and Tolerability of Talsaclidine in Patients With Mild to Moderate Dementia of the Alzheimer Type
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 506.208
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — talsaclidine fumarate

ARMS (1):
- Alzheimer (Experimental)
  Interventions: Drug: Talsaclidine

INTERVENTIONS:
Drug: Talsaclidine

SUMMARY:
Safety and tolerability. Quality of life (EQ-5D, ACQLI) and health economic impact (health resource utilisation, living and employment status) assessments, will not be performed at the centers in the united kingdom (UK)

ELIGIBILITY:
Inclusion Criteria:

* Patient met the inclusion criteria for the preceding talsaclidine trial
* Patient completed the preceding talsaclidine trial within the last four weeks with adequate compliance
* Patient is able to understand the patient information and give written informed consent in accordance with GCP (good clinical practice) and local legislation. In case of doubt, a study independent physician should assess the patient. If in the opinion of study independent physician the patient is unable to provide written inform consent, a legal guardian may provide consent on behalf of the patient
* Patient has a relative or caregiver who has given written informed consent to provide trial related information for self and patient and is willing and capable of supporting the clinical trial
* Patient and caregiver are able to complete the trial examinations, to hear, speak, read and write in a basic way and primary sensorial function are intact

Exclusion Criteria:

* Patient developed a medical condition during the preceding talsaclidine trial which, in the opinion of the investigator may be worsened by participation in this trial
* Patient experienced any serious drug related adverse event (s) in the preceding talsaclidine trial
* Patient dropped out of the preceding talsaclidine trial
* Patient was a major protocol violator in the preceding talsaclidine trial
* Untreated or non-compensated hypertension (BP systolic > 180 and/or diastolic > 110 mmHg)
* Hypertension being treated with ß-blockers
* Severe heart failure (NYHA: III and IV)
* Any arrhythmias including bradycardia with a rate of <50 bpm, arrhythmias due to second or third degree blocks and low II-IV, ECG <30 ventricular extra systoles/hour, multifocal or multiform and repetitive forms of ventricular extra systoles
* Bronchial asthma with phases of exacerbation or inducible by aspirin or other NSAIDSs
* Any patient with diabetes, type I or II, under active treatment with either insulin or any oral agent
* Renal insufficiency: calculated creatinine clearance below normal range (based on gender, age and weight)
* Acute hepatic disorder (liver enzymes above 50% upper normal limit)
* Patient has obvious symptoms of dehydration
* Neoplasm currently active or likely to recur (except basal cell carcinoma, squamous cell carcinoma of the skin and clinically significant meningioma)
* Patient is participating in another clinical trial
* Pregnant and lactating women, women of childbearing potential not using an approved method of contraception
* Insufficient compliance: in the investigator's opinion the patient or caregiver are unable to comply with the protocol requirements
* Exclude subjects with less than 50 kg body weight and/or with a calculated creatinine clearance below 50 ml/min. (It will be calculated by the central laboratory - values below normal range will be flagged by the central laboratory)
* Patients with abnormal urinalysis results such as infection or proteinuria as defined by:

  * A positive urinary bacterial culture, equal or greater than 10exp5 colony forming unit (CFU)/ml or
  * More than 10 leukocytes per high power field and with more than > 2 granular casts per low power field or
  * More than 10 red blood cells per high power field or
  * >+1 proteinuria (equivalent to >30 mg/dl) and with a ratio of urine protein/urine creatinine >0.3
* Any patient with a history of chronic urinary tract infection or recent urinary tract infection over the past six months. If the patient developed a lower urinary tract infection during their participation in the study 506.203 without any sign of kidney failure, then they are allowed to enter the study. Patients may continue in the trial only if the infection is confined to the lower urinary tract and without any sign of kidney failure, but must be discontinued otherwise
* Patients with a history of renal stones within the past six months

Concomitant Therapy exclusion

* Benzodiazepines (brotizolam, oxazepam, temazepam, or triazolam are allowed)
* Antidepressants including all tricyclics (trazodone is allowed; for clinically relevant depressed mood the Selective Serotonine Re-uptake Inhibitors (SSRIs) fluoxetine or paroxetine or sertraline are allowed)
* Antipsychotics (haloperidol or risperidone are allowed)
* Anticholinergics (topical application and promethazine is allowed)
* Lithium
* Acetylcholinesterase inhibitors
* Monoamine oxidase inhibitors
* ß blockers including topical application
* Any concomitant therapy with significant nephrotoxic potential in case of urinary tract infection (e.g. aminoglycoside, antibiotics and/or radiographic contrast agents)
* Hypericum perforatum (St John's wort) is excluded
* Use of neuroleptics within the trial: If the use of any neuroleptic is required during the course of the trial, the reason should be documented as an adverse event and the use of such medication should be limited. Use of neuroleptics should be stopped as soon as the patient's clinical status allows this to happen
* Patients receiving cognitive training prior to study entry are not excluded, but the training should be continued, if possible, throughout the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 1999-05; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 17 month after first drug administration
Number of patients with abnormal changes in laboratory tests | Up to 17 month after first drug administration

SECONDARY OUTCOMES:
Changes in neuropsychiatric inventory scores | Up to 17 month after first drug administration
Changes in clinical global impression (CGI)/ clinical global impression of change scores | Up to 17 month after first drug administration
Changes in mini mental state scores | Up to 17 month after first drug administration
Changes in quality of life by EuroQol (EQ-5D) score | Up to 17 month after first drug administration
  not to be performed in the United Kingdom
Assessment of healthy economic impact by healthy resource utilisation, living and employment status changes | Up to 17 month after first drug administration
  not to be performed in the United Kingdom
Changes in Alzheimer carer quality of life instrument (ACQLI) scores | Up to 17 month after first drug administration